CLINICAL TRIAL: NCT01142284
Title: Evaluation of Concomitant Administration of Cilostazol and Probucol on Biomarkers, Endothelial Function and Safety in Peripheral Artery Disease Subjects Complicated With Coronary Artery Disease.
Brief Title: Evaluation of Concomitant Administration of Cilostazol and Probucol on Biomarkers, Endothelial Function and Safety
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 021-KOA-0901i
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Peripheral Artery Disease
Keywords: Biomarker; Endothelial Function; Peripheral Artery Disease; Coronary Artery Disease; Flow Mediated Dilation; Cilostazol; Probucol
MeSH Terms: conditions — Peripheral Arterial Disease; Coronary Artery Disease | interventions — Cilostazol; Probucol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Cilostazol, Probucol
- Cilostazol (Experimental): cilostazol
  Interventions: Drug: Cilostazol, Probucol
- Probucol (Experimental): probucol
  Interventions: Drug: Cilostazol, Probucol
- Cilostazol + Probucol (Experimental): cilostazol and probucol
  Interventions: Drug: Cilostazol, Probucol

INTERVENTIONS:
Drug: Cilostazol, Probucol — Treatment Group 1 (control) No cilostazol or probucol
  Treatment Group 2 (cilostazol alone) 1 tablet cilostazol 100 mg PO BID
  Treatment Group 3 (probucol alone) 1 tablet probucol 250 mg PO BID
  Treatment Group 4 (concomitant cilostazol and probucol) 1 tablet cilostazol 100 mg PO BID, and 1 tablet probucol 250 mg PO BID

SUMMARY:
Based upon evidence of efficacy and safety of both cilostazol and probucol administration in independent randomized controlled trials in PAD and CAD, the present trial seeks to investigate the effect of concomitant administration of cilostazol and probucol on FMD compared to each drug individually, as well as to evaluate biomarker measures and safety indices in this context.

DETAILED DESCRIPTION:
Primary:

1. To evaluate the effect of concomitant administration of cilostazol and probucol on the 12-week change in FMD from baseline compared, with individual drugs alone.
2. To assess the safety of concomitant administration of cilostazol and probucol in peripheral artery disease (PAD) subjects complicated with coronary artery disease (CAD) as determined by physical examination, vital signs, adverse events (AEs), laboratory tests, ECGs.

Secondary:

1. To evaluate the effect of cilostazol and probucol administered concomitantly and as individual drugs, compared with control, on changes in FMD from baseline to Weeks 6 and 12.
2. To evaluate the effect of cilostazol and probucol administered concomitantly and as individual drugs, compared with control, on changes in metabolic, inflammatory, oxidative, and platelet biomarkers from baseline to Weeks 6 and 12.
3. To evaluate the effect of cilostazol and probucol administered concomitantly and as individual drugs, compared with control, on the time course (over the 12-week treatment period) of changes in FMD and biomarkers levels.
4. To assess the effect of drug withdrawal on these endpoints at follow-up (from Week 12 to Week 16).
5. To explore the relationship between changes in FMD and changes in the biomarker levels at Week 12.

ELIGIBILITY:
Inclusion Criteria:

1. Age is ≥ 40 and <80 years at Screening.
2. The subject has a diagnosis of PAD
3. The subject has a diagnosis of CAD
4. Stable background medical therapy over the past 3 months
5. Taking 100mg/day of aspirin or 75mg/day of clopidogrel over the past 3 months
6. Hyperlipidemia defined as a LDL cholesterol concentration > 70 mg/dL
7. The subject is willing to participate in this study as documented by written informed consent

Exclusion Criteria:

1. New diagnosis of PAD within 3 months.
2. Currently taking cilostazol or has taken cilostazol
3. Currently taking probucol or has taken probucol within the last 3 months
4. Critical limb ischemia (CLI)
5. Congestive heart failure
6. Transient ischemic attack (TIA)
7. Endovascular peripheral or coronary revascularization procedure within 3 months
8. Coronary artery bypass graft (CABG) or major cardiovascular surgical procedures within 6 months
9. Major surgical procedures within 3 months
10. Uncontrolled hypertension
11. Type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus
12. Diabetic complications of severe peripheral neuropathy or active retinopathy.
13. Inflammatory bowel disease.
14. Unstable angina
15. QT prolongation
16. Severe or life threatening ventricular arrhythmias
17. History of syncope
18. Serum creatinine > 2.5 mg/dL, Creatinine Clearance ≤25ml/min or renal failure requiring dialysis.
19. History or evidence of any hematological or clotting disorder.
20. Hematocrit ≤ 28% or ≥ 55%.
21. AST or ALT > 3 times the upper limit of normal (ULN).
22. Any form of chronic anticoagulation.
23. Coagulopathies defined as an INR > 1.5
24. History of malignant disease within 5 years.
25. Acute or chronic hepatitis.
26. Hemophilia or known increased risk of hemorrhage.
27. Other clinically significant disorders resulting in a remaining life expectancy less than one year.
28. Current alcohol or drug abuse.
29. If female, the subject cannot be pregnant or breastfeeding and must be of non-childbearing potential

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2012-11-29 (Actual); Study Completion 2012-12-18 (Actual)

PRIMARY OUTCOMES:
On the 12-week change in FMD / Safety | 12 weeks
  1. To evaluate the effect of concomitant administration of cilostazol and probucol on the 12-week change
  2. To assess the safety of concomitant administration of cilostazol and probucol

SECONDARY OUTCOMES:
Changes in the biomarker and FMD | 12 weeks
  1. To evaluate the effect of cilostazol and probucol administered concomitantly and as individual drugs, compared with control, on changes in FMD
  2. To evaluate the effect of cilostazol and probucol administered concomitantly and as individual drugs, compared with control on biomarkers
  3. To evaluate the effect of cilostazol and probucol administered concomitantly and as individual drugs, compared with control, on the time course
  4. To assess the effect of drug withdrawal
  5. To explore the relationship between changes in FMD and changes in the biomarker levels

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea